CLINICAL TRIAL: NCT03192761
Title: The Best Method for ACL Reconstruction. A Study Comparing Reconstructions of Anterior Cruciate Ligament Using Grafts Taken From Three Different Anatomical Locations at the Knee and Thigh. A Randomized Clinical Trial
Brief Title: The Best Method for ACL Reconstruction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lars Konradsen (Other)
Responsible Party: Sponsor-Investigator, Lars Konradsen, Senior consultant, clinical professor, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BBH-ACL-1
Record Dates: First submitted 2017-04-27; First posted 2017-06-20 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Intervention Model Description: When the patient has been anaesthetized for surgery, the method of reconstruction is defined by opening a sealed envelope in the operating theatre.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessor is not involved in the surgical procedures. Participants wear long trousers at follow-up procedures to mask surgical incisions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACL-reconstruction hamstrings (Active Comparator): ACL reconstruction hamstrings
  Interventions: Procedure: ACL reconstruction hamstrings
- ACL-reconstruction patella tendon (Active Comparator): ACL reconstruction patella tendon
  Interventions: Procedure: ACL reconstruction patella tendon
- ACL-reconstruction iliotibial tract (Active Comparator): ACL reconstruction iliotibial tract
  Interventions: Procedure: ACL reconstruction iliotibial tract

INTERVENTIONS:
Procedure: ACL reconstruction hamstrings — HG reconstruction is performed according to the standard procedure of the department:
  A double semi-Tendinosus and gracillis graft is used. Placement of the bony tunnels is anatomical, and the femoral tunnel is positioned through the antero-medial portal. Fixation proximally is by CL-endobutton and at the tibia by Intrafix sheet and screw
  Arms: ACL-reconstruction hamstrings
Procedure: ACL reconstruction patella tendon — PTBG reconstruction is performed according to the standard procedure of the department:
  A bone patella tendon bone graft of 1 cm width from the midportion of the tendon is used. Placement of the bony tunnels is anatomical, the femoral being positioned through the antero-medial portal. Fixation proximally and distally is by interference screws.
  Arms: ACL-reconstruction patella tendon
Procedure: ACL reconstruction iliotibial tract — TIFLG reconstruction is performed as follows:
  The TIFL graft is harvested using two lateral incisions. The graft is left attached to the distal iliotibial tract. Placement of the bony tunnels is anatomical, the femoral being drilled outside-in. The tibial drill tunnel is made by retrograde drilling 20 mm, leaving cortical bone at the distal end of the tunnel. Fixation distally is by CL-endobutton or interference screw and on femur by an interference screw outside-in.
  Arms: ACL-reconstruction iliotibial tract

SUMMARY:
The investigators wish to compare 3 methods for reconstruction of the anterior cruciate ligament using 3 different grafts: bone-patella tendon-bone, hamstrings and iliotibial tract graft, as these methods influence the muscles around the knee differently. Methods using bone-patella tendon-bone and hamstrings are performed as standard operations, and the use of the iliotibial tract graft using a new method of reconstruction.

The purpose is:

1. To assess whether one of three different grafts used for reconstruction of the ACL shows superior results compared to the others in relation to mechanical stability and re-rupture rates.
2. To assess whether one of three different methods for reconstruction of the ACL shows superior results compared to the others in subjective patient outcome measures.
3. To assess whether one of three different methods for reconstruction of the ACL shows superior results compared to the others when considering specific symptoms and complications that can be related to donor-site morbidity.
4. To assess whether one of three different methods for reconstruction of the ACL shows superior results compared to the others when considering muscular power, muscle coordination, and function.

DETAILED DESCRIPTION:
The purpose of the study is described in the "Brief Summary" section.

Patients scheduled for ACL reconstruction at the Section of Arthroscopic Surgery and Sports Traumatology M51, Department of Orthopedics, Bispebjerg-Frederiksberg Hospital are eligible for this study Eligibility criteria are described in the "Eligibility" section.

The patients are scheduled for ACL surgery at consultation with a doctor from the Section of Arthroscopic Surgery and Sports Traumatology after usual, clinical criteria. The doctor informs the patient about the project, gives the patient the written patient information, and if the patient shows interest in the study, an appointment is scheduled with one of the surgeons involved in the project.

At this appointment the patient is informed about the project by the surgeon. The patients will be granted the reflection time they need before consenting or rejecting.

Before the day of surgery muscle power, muscle coordination and functional tests are performed, and objective tests and PROMs are completed.

Surgery is performed by one of two surgeons experienced in all three methods of surgery as described in the "Arms and Interventions" section.

After the patient is put under general anaesthesia the method of ACL reconstruction is chosen by opening a sealed envelope.

Outcome measures are recorded at 1-year and 2-year follow-up.

All three methods of reconstruction are believed to have the same risk for basic complications: infection (approx. 1%), stiffening of the knee (approx. 2%) and deep venous thrombosis (approx. 1 %)

It is assumed that a 20% difference in a patient reported outcome score (KNEES-ACL) represents a clinically relevant difference. Based on standard deviations for the outcome score, and with a 90% power, significant differences of 20 % can be shown in a sample of 20 patients. Significance level is set at 5%. The investigators aim for 30 patients in each group, considering potential drop-outs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an ACL rupture scheduled for ACL reconstruction after clinical investigation by an orthopedic specialist at the Section of Sports Traumatology M51.
* Age 18-40 years.
* Patients able to understand given information in relation to the study and to complete out-come questionnaires.

Exclusion Criteria:

* Patient activity (sports or work) that excludes one or more of the three methods of surgery, e.g. work predominantly performed kneeling would exclude the use of the BPTBG.
* Other ligament injuries (except non-surgically treated lesion of MCL - medial collateral ligament) to the same knee or ligament injury (except non-surgically treated lesion of MCL - medial collateral ligament) to the contralateral knee
* Conditions in either knee with pain of such intensity, that participation in the functional tests of this study are impossible.
* Auto-immune disease that involves lower limb joints or muscles.
* Local or systemic infection.
* Actual or previous systemic corticosteroid, chemotherapeutic, or immunosuppressive treatment.
* BMI>30.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in KNEES-ACL score | pre-op, 1 year, 2 years
  patient-reported outcome measure

SECONDARY OUTCOMES:
Change in anterior-posterior stability (quantified by Rolimeter) | pre-op, 1 year, 2 years
  Measure of anterio-posterior laxity
Change in graded pivot shift | pre-op, 1 year, 2 years
  Subluxation of the tibia relative to the femur
Change in muscle strength and forward lunge ability | pre-op, 1 year, 2 years
  Result of muscle power and muscle coordination tests

CONTACTS AND LOCATIONS:
Overall Officials: Michael Krogsgaard, Study Director — Head of section
Locations (1):
- Bisppebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Yes